CLINICAL TRIAL: NCT03457961
Title: Post-market Study of AMPA Receptor Antagonists for Epilepsy Patients in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Howan Leung, Associate consultant, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: 2016-HL-001
Record Dates: First submitted 2018-02-25; First posted 2018-03-08 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Focal Epilepsy; Generalized Epilepsy; Partial Seizures, Simple
Keywords: Perampanel; focal onset seizure; epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy, Generalized; Seizures; Epilepsy | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adjunctive Perampanel: A group of patients who aged 12 years or above and have a diagnosis of epilepsy with simple partial seizure and/or complex partial seizures
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — This study collects clinical information during the first 16 weeks after the first dose of AMPA/NMDA receptor antagonist. Subjects or caregivers shall provide seizure diary which documents seizure type and seizure frequency as per usual medical care. The final visit will be based on the week-16 visit.
  Other Names: Fycompa

SUMMARY:
Background:

Epilepsy is a chronic neurological disease which affects approximately 70,000 patients in Hong Kong and 50 billion people worldwide. Among these patients one-third remained unresponsive to antiepileptic agents. Continual drug manipulation is an essential therapeutic option for these patients with refractory epilepsy. In particular, rational polytherapy has become the mainstay of treatment for the sub-group of patients who have failed two or more antiepileptic drugs (AEDs).

A substantial amount of research has shown that N-methyl-D-aspartate receptors (NMDA) may play a key role in the pathophysiology of several neurological diseases, including epilepsy. Animal models of epilepsy and clinical studies demonstrate that NMDA receptors activity and expression can be altered in association with epilepsy and particularly in some specific seizure types. NMDA receptor antagonists have been shown to have antiepileptic effects in both clinical and preclinical studies. There is some evidence that conventional antiepileptic drugs may also affect NMDA receptor function.

Aims:

To investigate the medium to long-term effects of AMPA/NMDA receptor antagonist in an Asian cohort as there is a relative lack of clinical data in this population To explore the efficacy of AMPA/NMDA receptor antagonist in patients with partial onsets seizures that may secondarily generalize and the specific side effects of AMPA/NMDA receptor antagonist in relation to behavioral problems.

Methods:

A semi-prospective design is adopted to recruit patients who are indicated and started on AMPA/NMDA receptor antagonist aged 12 or above in Hong Kong. This study will collect information about demographic details, medical history and seizure information. Assessment of seizure frequency is based on seizure diary and interviews with family members. Physical examination, electrocardiogram and other medical information relevant to the follow-up of the patient will be collected.

DETAILED DESCRIPTION:
Epilepsy is a chronic neurological disease which affects approximately 70,000 patients in Hong Kong and 50 billion people worldwide. Among these patients, one-third remained unresponsive to antiepileptic agents. Continual drug manipulation is an essential therapeutic option for these patients with refractory epilepsy. In particular, rational polytherapy has become the mainstay of treatment for the sub-group of patients who have failed two or more antiepileptic drugs (AEDs).

Using AEDs with different mechanisms of action is a strategy adopted by many doctors around the world. In this regard, perampanel (PER) is an agent which is first in its class, with specific antagonistic action on ionotropic α-amino-3-hydroxy-5-methyl-4-isoxazoleproprionic acid (AMPA) glutamate receptor of post-synaptic neurons. The pharmacokinetics of PER suggested that it has a half-life of approximately 105 hours and the steady-state concentrations that can be reached in 14 days. PER is approximately 95% bound to plasma proteins. This metabolism is mediated by CYP 3A4 or CYP 3A5. The usual dosage of PER is between 2mg and 12 mg. PER can be administered once daily.

A total of five clinical studies demonstrated the efficacy of PER among patients with refractory epilepsy. These were all double-blind studies and all of them evaluated the 50% responder rate as a seizure outcome. The corresponding risk ratio for 50% responder rates for 4mg, 8mg and 12mg were 1.54, 1.8 and 1.72. The most common treatment-emergent adverse effects were dizziness, drowsiness, headache, fatigue, nasopharyngitis. The pooled results suggested that a higher dose was more efficacious if the side effects could be tolerated. There was an on-going study on the use of PER among patients with secondarily generalized seizures. Perampanel has been approved in many countries such as USA, EU, Australia, Canada, Switzerland, Singapore, and Malaysia, as an adjunctive therapy for refractory partial seizures with or without secondary generalisation among patients above 12 years of age.

A substantial amount of research has shown that N-methyl-D-aspartate receptors (NMDA) may play a key role in the pathophysiology of several neurological diseases, including epilepsy. Animal models of epilepsy and clinical studies demonstrate that NMDA receptors activity and expression can be altered in association with epilepsy and particularly in some specific seizure types. NMDA receptor antagonists have been shown to have antiepileptic effects in both clinical and preclinical studies. There is some evidence that conventional antiepileptic drugs may also affect NMDA receptor function.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged 12 years or above
2. Subject has a diagnosis of epilepsy with simple partial seizure and/or complex partial seizures
3. Subjects who have a baseline seizure rate of more than 2 per month in the eight week period preceding the start of AMPA / NMDA receptor antagonist
4. No seizure free period longer than 21 days during the eight week period before AMPA receptor antagonist was started
5. Patients who already had neuropsychiatric inventory completed twice during the treatment period spanning at least 16 weeks.

Exclusion Criteria:

1. Subjects with idiopathic generalised epilepsy (for example, juvenile myoclonic epilepsy and absence epilepsy)
2. Patients who only suffer from isolated auras
3. Baseline creatinine clearance of less than 50ml/min
4. Severe hepatic impairment with ALT three times the upper limits of normal
5. Significant psychiatric conditions before the start of AMPA / NMDA receptor antagonist
6. Progressive neurodegenerative conditions
7. Active history of malignancy
8. History of severe haematological conditions or serious blood dyscrasias
9. Corrected QT interval more than 450 milli-second on ECG
10. Substance abuse
11. Pregnancy, breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (diagnosed epilepsy with simple partial seizure) who have a baseline seizure rate of more than 2 months would be provided perampanel as adjunctive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-07-23 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy end-points | 16 weeks
  The primary efficacy end-points evaluates seizure frequency (per month) in week 0 (baseline) and week 16 (maintenance phase). The investigators will used those seizure frequencies (per month) to calculate the percentage change from baseline to maintenance phase for each subject and categories: no change, between 0 to 50% decrease, 50% to 75% decrease, 75% to 100% decrease.
Seizure freedom rate in study population | 16 weeks
  The proportion of subjects achieving seizure freedom during the maintenance period will be documented. The percentage of seizure free days in the maintenance phase will also be collected. The investigators will report the seizure freedom rate for the present study population and the average days of achieving seizure freedom.

SECONDARY OUTCOMES:
Psychiatric and behavioral adverse events | 16 weeks
  The investigators would use the Neuropsychiatric Inventory Questionnaire (NPI) with 12 domains to evaluate the neuropsychiatric events in week 0 (baseline) and week 16 (maintenance phase). The investigators will record each symptom severity (rated 1 occasional to 4 very frequent) and frequency (rated 1 mild to 3 severe).

CONTACTS AND LOCATIONS:
Overall Officials: Ho Wan Leung, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
This is a cohort study for perampanel in Hong Kong. There is no plan to make individual participant data to share. The results would be shared in publications. Electronic data will be saved in secured computer of the individual sites with restricted access. The anonymous data will be managed installed for developing future studies.

REFERENCES:
- [Background] Steinhoff BJ, Bacher M, Bast T, Kornmeier R, Kurth C, Scholly J, Staack AM, Wisniewski I. First clinical experiences with perampanel--the Kork experience in 74 patients. Epilepsia. 2014 Jan;55 Suppl 1:16-8. doi: 10.1111/epi.12492. PMID 24400693
- [Background] Juhl S, Rubboli G. Perampanel as add-on treatment in refractory focal epilepsy. The Dianalund experience. Acta Neurol Scand. 2016 Nov;134(5):374-377. doi: 10.1111/ane.12558. Epub 2016 Jan 13. PMID 26763771
- [Background] Trinka E, Steinhoff BJ, Nikanorova M, Brodie MJ. Perampanel for focal epilepsy: insights from early clinical experience. Acta Neurol Scand. 2016 Mar;133(3):160-72. doi: 10.1111/ane.12529. Epub 2015 Oct 28. PMID 26506904